CLINICAL TRIAL: NCT01247688
Title: Umbilical Cord Blood Transplant for Children With Lymphoid Hematological Malignancies (UCALL)
Brief Title: Umbilical Cord Blood Transplant for Children With Lymphoid Hematological Malignancies
Acronym: UCALL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn due to low accrual.
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Caridad Martinez, Assistant Professor, Pediatric Hematology/Oncology, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26336-UCALL
Record Dates: First submitted 2010-11-17; First posted 2010-11-24 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoid Hematological Malignancies; Umbilical Cord Blood Transplant
Keywords: Lymphoid; hematologic malignancy; UCB; Umbilical Cord Blood Transplant; Total Body Irradiation; Cytoxan; Cyclophosphamide; Fludarabine
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical Cord Blood Transplant Treatment Plan (Experimental): Cytoxan, Fludarabine, Total Body Irradiation (TBI), Cord Blood Stem Cell Infusion
  Interventions: Drug: Cytoxan; Drug: Fludarabine; Radiation: Total Body Irradiation (TBI); Procedure: Cord Blood Stem Cell Infusion

INTERVENTIONS:
Drug: Cytoxan — 50 mg/kg/dose will be given IV on day -5,-4, -3, -2 over 1 hour. The total dose to be given over 4 days is 200 mg/kg.
  Other Names: Cyclophophamide
Drug: Fludarabine — 40mg/m2/day will be given IV over 1 hour on day -4, -3, -2
  Other Names: Fludara
Radiation: Total Body Irradiation (TBI) — 1.75Gy/fraction will be given on day -9, -8, -7, -6
Procedure: Cord Blood Stem Cell Infusion — The cord blood stem cells will be infused on day 0

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of UCBT to treat patients with lymphoid hematological diseases and to see if this treatment can decrease the incidence of leukemia relapse, GVHD and infections.

These patients have a type of blood cell disorder that is very hard to cure. This treatment that is being used in this trial is known as a stem cell transplant. This treatment might help the patient live longer without the disease. It uses much stronger doses of drugs and radiation to kill the diseased cells that could be given without the transplant. We also think that the healthy cells from the donor may help fight any diseased cells left after the transplant.

For the transplant to take place, we will administer stem cells from a 'donor' whose cells best 'match' the patient's. In this study umbilical cords will be the source of the stem cells. Before the transplant, two very strong drugs plus total body irradiation will be given to as preconditioning. This treatment will kill most of your blood-forming cells in the bone marrow. The patient will then get then healthy stem cells.

If the patient has the disease in the central nervous system (CNS), they will receive radiation to the head and spine before starting the conditioning. This is to try to get disease control in the CNS. Radiation will not be given for children under 2 yrs old.

Currently, many umbilical cord blood units are available in public banks for transplantation in patients lacking bone marrow donors. UCB transplants (UCBT) may offer several advantages over adult bone marrow or peripheral blood stem cell transplants, including:

1. rapid availability,
2. absence of donor risk,
3. low risk of transmissible infectious diseases,
4. low risk of acute GvHD (Graft vs. Host Disease)

The three main causes of death after umbilical cord blood transplantation for these kind of disorders are graft failure, infection and disease relapse.

In this study we are trying to address these three problems:

To help improve engraftment we will add the drug Fludarabine to Cytoxan and total body irradiation. Fludarabine is a very strong medicine. We will try to decrease infections and reduce leukemia relapse by using fludarabine instead of antithymocyte globulin (ATG).

DETAILED DESCRIPTION:
After the eligible criterion for treatment has been met and a suitable UCB stem donor has been found, the patient will have a central line placed.

Research Therapy:

After placement of the central line, the following chemotherapy will be given to after admission to the hospital and before the infusion of the umbilical cord blood stem cells:

* 9 - 6 days before the infusion: Total Body Irradiation (TBI) in two fractions ("doses") per days.
* 5 - 2 days before the infusion: Cytoxan given daily for 4 days, over 1 hour as an intravenous infusion. Mesna will be given per standards. Mesna is a drug given to decrease the side effects of Cytoxan. It will be given daily as an intravenous infusion while the patient receives the Cytoxan.
* 4 - 2 days before the infusion: Fludarabine given daily for 3 days over 1 hour as an intravenous infusion.

Stem cell transplant (intravenous infusion of the UCB stem cells) - defined as day 0 of the treatment. All other "numbered" days relate to this infusion date. For example, Day 1 is the first day after the stem cell transplant.

The following medications will be given to help decrease side effects from the chemotherapy and UCB infusion: Cyclosporine A (CSA) will be given starting 3 days prior to the stem cell infusion. It will be given daily over 2 hours every 12 hours, after the infusion and then tapered if no GVHD is present.

Administration of Mycophenolate mofetil (MMF) will start on the day the stem cell infusion is completed and will continue daily for 45 days, unless the patient develops GvHD.

Intravenous immunoglobulin's (IVIG) will be given monthly until GVHD therapy is stopped and there is evidence that the patient's body is producing antibodies.

Study Evaluations: Various study evaluations will be performed before and during the trial.

Follow Up: After year 1, the patient will be asked to return to the clinic once a year for consultations and bone marrow tests. A follow up bone marrow biopsy and aspirate will be done 1 and 2 years after transplant. Consultations with specialists will be similar to the ones the patient had before the transplant.

ELIGIBILITY:
INCLUSION CRITERIA:

* Potential recipients of umbilical cord blood transplantation (i.e. HLA (human leukocyte antigen) matched or mismatched / related or unrelated) with a lymphoid hematologic malignancy (acute lymphoblastic leukemia, hodgkin/non-hodgkin lymphoma) unlikely to be cure by standard chemotherapy. This includes patients who have relapsed after standard chemotherapy treatments and patients in first remission with unfavorable prognostics features.
* Related or Unrelated Umbilical Cord Blood Unit with 0-1 antigen mismatch, Total Nucleated cell dose of greater than or equal to 4 x 10^7/kg.
* Lansky/Karnofsky scores greater than or equal to 60
* Negative pregnancy test (if applicable)
* Written informed consent and/or signed assent line from patient, parent or guardian.

EXCLUSION CRITERIA:

* Patients with uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic antifungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Severe renal disease (Creatinine > x 3 normal for age)
* Severe hepatic disease (direct bilirubin > 3 mg/dl or SGOT (Serum glutamic oxaloacetic transaminase) > 500)
* Patient has DLCO (Diffusing Capacity of the Lung for Carbon Monoxide) < 50% predicted or FEV1 (Forced expiratory volume ) < 50% of predicted, if applicable
* Patients with symptomatic cardiac failure unrelieved by medical therapy or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction<20%).
* HIV positive

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival at 1 year after UCB transplant in pediatric patients | 1 year
  To determine the survival rate at 1 year after umbilical cord blood transplant in pediatric patients with lymphoid hematological malignancies

SECONDARY OUTCOMES:
Assessment of Platelet Count Recovery | Day 42
  To assess platelet recovery at day 42 post transplant
Number of participants with severe acute GVHD grade III-IV as an assessment of safety | Day 100
  To estimate the risk of severe grade III-IV acute GvHD at day 100.
Number of participants with chronic GvHD as an assessment of safety | 1 year
  To estimate the risk of chronic GvHD at 1 year
Assess relapse rate after transplant | 1 and 3 years
  To assess relapse rate at 1 and 3 years after transplant.
Assessment of neutrophil count recovery | Day 42
  To assess neutrophil count recovery at day 42 post transplant
To evaluate cell recovery and function | day 100, 6, 12, and 24 months
  To evaluate T/B/NK cell recovery and function at day 100, 6, 12, and 24 months after transplant.
Assess leukemia free survival | 1 and 3 years
  To assess leukemia free survival at 1 and 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Caridad A Martinez, MD, Principal Investigator — Baylor College of Medicine; Robert A Krance, MD, Principal Investigator — Baylor College of Medicine